CLINICAL TRIAL: NCT04815499
Title: Study of the Impact on Quality of Life With ARACOMPLEX® Food Supplement Versus Placebo in Chronic Obstructive Pulmonary Disease Patients With a CAT Score> 15.
Brief Title: Effects of a Food Supplement on Quality of Life in Patients With Chronic Obstructive Pulmonary Disease.
Acronym: EPOCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arafarma Group, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ARA-EXP/ARA-2019-01
Record Dates: First submitted 2021-01-28; First posted 2021-03-25 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food supplement (Experimental): One tablet a day, during 12 months
  Interventions: Dietary Supplement: Food supplement
- Placebo (Placebo Comparator): One tablet a day, during 12 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Food supplement — ARACOMPLEX® is an authorized food supplement that contains maca extract, vitamin complexes and ions, and that improves the quality of life of the patient.
  Arms: Food supplement
Dietary Supplement: Placebo — Placebo has a composition that makes its weight and organoleptic characteristics are identical to ARACOMPLEX®.
  Arms: Placebo

SUMMARY:
It has been demonstrated that consequences of malnutrition affect a situation of risk and have negative effects on the evolution of chronic obstructive pulmonary disease (COPD), accompanied by higher morbidity and mortality. The impact of malnutrition on the respiratory system affects the respiratory muscles, the lung parenchyma, and the immune system. In summary, the risk of complications can lead to a worsening of the quality of life of the COPD patient. Also, dyspnea as the main symptom of COPD is the one that produces the greatest loss of quality of life, especially in older patients. The components of our authorized food supplement improve the quality of life of the patient. These components maintain the strength and energy of the patient, help the body to recover and regain its optimal state, help improve the immune system, help reduce the side effects of therapies associated with the control or cure of cancer and help correct nutritional deficiencies. This is the reason why this experimental study aims to improve the quality of life in patients with COPD with a CAT score>15.

DETAILED DESCRIPTION:
This study is developed in two phases: pilot phase and experimental phase. The pilot phase is preliminary and progressive in order to demonstrate a sufficient effect of improving the quality of life of patients and to be able to continue in an experimental phase with more investigational sites and more patients, and to evaluate other secondary objectives.

Once the pilot phase is finished, an intermediate analysis of the results will be carried out to evaluate the magnitude of the variation in quality of life at 3, 6, 9 and 12 months. If the expected success expectations are achieved and it is approved by the Ethics Committee, the study will continue to the experimental phase.

ELIGIBILITY:
Inclusion Criteria:

* Adults: men and women ≥ 18 years.
* Patients with a medical diagnosis of COPD based on a recent spirometry.
* Patients with a CAT score> 15, affecting COPD symptoms in a moderate-high way in the daily life of these patients.
* Minimum clinical stability period of 4 weeks before the start of the study.
* Patients who are trained to give informed consent.
* Patients must agree to perform study visits and procedures with precise instructions.

Exclusion Criteria:

* BMI ≥ 40.
* Comorbidities, which due to their severity or progression, may interfere with the results, such as cancer, hematological disorders, severe heart or liver failure, kidney failure on dialysis, tuberculosis (TB) or AIDS, or other pulmonary pathologies such as pulmonary thromboembolism ( PE), pulmonary fibrosis, or relevant bronchiectasis.
* In Pulmonary Rehabilitation treatment or in treatment for smoking.
* Pregnancy or breastfeeding.
* Impossibility of the patient, due to a medical condition, to follow the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | 12 months
  To assess the magnitude of the change from baseline quality of life at 3 months, 6 months, 9 months and 12 months using the COPD Assessment Test (CAT) scale in COPD patients with a CAT score> 15 who receive ARACOMPLEX® supplementation compared to those patients receiving placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Doctor Peset, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided